CLINICAL TRIAL: NCT04344470
Title: Study of Volition: Behavioral Analysis and Clinical Neurophysiological Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200077; 20-N-0077
Record Dates: First submitted 2020-04-11; First posted 2020-04-14 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03-21

CONDITIONS: Normal Physiology
Keywords: Healthy Volunteers
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Healthy Volunteers
  Interventions: Device: EMG; Device: EEG

INTERVENTIONS:
Device: EMG — EMG will be recorded from two electrodes placed on both extensor carpi radialis (ECR) muscles
Device: EEG — EEG electrodes will be positioned according to 10-20 International System, with every impedance kept under 5 kOhm. EEG data will be amplified, filtered (DC-100 Hz), digitized at 1000 Hz, and stored on a computer for offline analysis.

SUMMARY:
Background:

'Free will' can be defined as the belief that people have control over their thoughts and movements. The topic of free will is controversial and is still being debated. Science has only partial answers to questions about free will, so researchers want to learn more about it. They want to assess the role of consciousness when intentions are present with behavior. This could help to explain the causal role of consciousness in movement or decisions.

Objective:

To learn more about free will.

Eligibility:

Healthy, right-handed adults ages 25-45

Design:

Participants will be screened with medical history, physical exam, and neurological exam.

Participants will have 1 study visit. It will last up to 4 hours.

Participants will sit in a comfortable chair in front of a screen. They will perform some or all of the following tasks.

Visual Task. Participants will watch different stimuli on the screen and answer simple questions.

Electroencephalography (EEG). An EEG records the electrical activity of the brain ('brain waves'). For the EEG, small electrodes are put on the scalp with an electrode cap. A gel is placed in the space between the electrodes and the scalp. Participants' brain waves will be recorded, including while they decide whether to move their thumb.

Choice/Reaction Time Task. Participants will watch different stimuli on the screen and react to them by moving their wrist. During this task, they will wear an EEG cap on their head and electrodes on their arms and wrists.

Electromyography. Small electrodes will be attached to participants' skin. Their muscle activity will be recorded while they decide whether to move their wrist and during the movement itself.

Transcranial Magnetic Stimulation (TMS): TMS is a non-invasive brain stimulation that uses magnetic field to stimulate nerve cells in your brain. TMS can increase or decrease brain activity in particular area of your brain. TMS operates completely outside of the body and is generally very well tolerated....

DETAILED DESCRIPTION:
Study Description:

The main focus of this protocol will be to try to identify the quale of free will, its electrophysiological correlates, and to determine whether this quale plays a causative role in movement.

Objectives:

Primary Objectives:

We will be doing a series of experiments. In the first experiments, we want to explore the behavioral response of normal subjects when they move after a visual stimulus that can be seen or unseen. We want to study behavior in different conditions with movement triggered by stimuli that are seen and not seen. Furthermore, we want to analyze the EEG related to those stimuli to explore sensory and motor processing.

Endpoints:

Primary Endpoints:

Reaction time and accuracies of the responses to different stimuli in different conditions will be identified as well as the subjects subjective experiences. EEG ERP shapes and microstates patterns will also be investigated.

Study Population:

Up to 50 healthy volunteers of both genders between the ages of 25-45, fluent in English and right-handed.

Participant Duration:

The total study is expected to last 48 months, with each individual expected to participate in a single 4-hour outpatient visit at the NIH Clinical Center, but there can be multiple visits.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Age between 25-45 years
* Right-handed (tested by the Edinburg handedness inventory).
* Able to give informed consent.
* Able to comply with all study procedures.
* Fluent in English.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Illegal drug use within the past 6 months based on history alone. The intent is to exclude those with drug use that may affect study results.
* Self-reported consumption of >14 alcoholic drinks/week for a man and >7 alcoholic drinks/week for a woman.
* Abnormal findings on neurological examination.
* History of current brain tumor, stroke, head trauma with loss of consciousness, epilepsy, or seizures.
* Current episode of major depression or any major psychiatric illness.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Experiment1: Identification of the best characteristics that allow us to create a backward masking effect of the second stimulus on the first one. | throughout
  We will develop a methodological approach to create the best backward masking effect. We will ask the subjects what they saw, to prove the effectiveness of the backward masking.
Experiment 2: Reaction time and accuracies of the responses to different stimuli (symbols, faces, objects, etc.) in different conditions (with and without masking) | throughout
  Subjects will move to the first stimulus even if unseen. We want to study subjects behavior in different conditions (simple reaction task, choice reaction task, with and without masking) with different stimuli (symbols, faces, objects, etc.). Furthermore, we want to analyze the EEG (classic ERP, microstates, etc.) related to those stimuli. EEG will be also analyzed to study the nature and strength of the visual pathway for movement and the pathway for visual perception at rest.
Experiment 1: Identification of the EEG characteristic or ERP shape related to different stimuli and the brain region origin. | throughout
  We will create a template of the shape of the ERP and the characteristics of EEG related to different stimuli to be identified in the second sub-study.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren B Reoma, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
.This will be determined at a later time. It is not yet known if it is feasible to share IPD.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-N-0077.html